CLINICAL TRIAL: NCT06867172
Title: The Emerging Issue - Pancreatic Steatosis Prevalence in Pancreatic Cystic Neoplasms and Adenocarcinoma: Insights From a Single-center Retrospective Study
Brief Title: Prevalence of Pancreatic Steatosis in Pancreatic Cystic Neoplasms and Pancreatic Adenocarcinoma
Acronym: SPACE
Status: Recruiting | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Vladut Catalina, Principal Investigator, Gastroenterologist, Assistant Lecturer University of Medicine and Pharmacy, Carol Davila University of Medicine and Pharmacy
Other Study IDs: 346833
Record Dates: First submitted 2024-09-27; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Steatosis; Pancreatic Cyst; Pancreatic Adenocarcinoma
Keywords: pancreas; steatosis; cyst; cancer; adenocarcinoma; fat
MeSH Terms: conditions — Pancreatic Cyst; Fatty Liver; Cysts; Neoplasms; Adenocarcinoma; Platelet Glycoprotein IV Deficiency | interventions — Tomography, X-Ray Computed; Endosonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pancreatic cyst: Neoplastic pancreatic cystic lesion
  Interventions: Diagnostic Test: computerized tomography; Diagnostic Test: Endosonography (EUS)
- PDAC: Pancreatic ductal adenocarcinoma for supplementary analysis
- Control group: Control group for comparison

INTERVENTIONS:
Diagnostic Test: computerized tomography — Little is known about the prevalence of pancreatic steatosis in patients with pancreatic cystic lesions therefore this observational study aims to clarify the data.
  Groups: Pancreatic cyst
Diagnostic Test: Endosonography (EUS) — EUS can better evaluate all pancreatic cysts, therefore is mandatory in this observational study.
  Groups: Pancreatic cyst

SUMMARY:
Several pancreatic neoplastic cystic lesions, such as IPMN (intrapapilary mucinous neoplasia), cystic neuroendocrine tumors (NET) and mucinous neoplasms, present a carcinogenetic risk, though it is yet unknown if this risk is increased in patients with pancreatic steatosis (PS).

The primary objective of the study is to determine de prevalence of pancreatic steatosis in pancreatic neoplastic cysts and if pancreatic steatosis is increased in those lesions that pose a carcinogenetic risk.

The secondary objective is to evaluate the prevalence of pancreatic steatosis in pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic steatosis has gained significant novel interest in the pathophysiology of PDAC and neoplastic cystic lesions. Pancreatic steatosis is the new emerging issue in pancreatology. Recently, pancreatic steatosis has gained significant novel interest in the pathophysiology of PDAC.

The primary objective of the study is to determine de prevalence of pancreatic steatosis in pancreatic neoplastic cysts and if pancreatic steatosis is increased in those lesions that pose a carcinogenetic risk.

Pancreatic ductal adenocarcinoma (PDAC) has a poor survival, predominantly as a result of its diagnosis in advanced stages. Pathological changes of steatosis are an independent determinant of PDAC, and these pathological changes are correlated with the attenuation of the pancreas on computed tomography (CT). The secondary objective is to evaluate the prevalence of pancreatic steatosis in pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patients with at least 1 pancreatic cystic lesion based on CT and EUS features, with a cyst size ≥ 5mm; or healthy subjects or PDAC (confirmed by histopathological exam).

Exclusion Criteria:

* No evidence of written informed consent
* Patients with contraindications for endoscopy due to comorbidities
* Metal stent in hepato-bilio-pancreatic region at time of baseline CT-imaging (vascular, luminal and biliary)
* Acute pancreatitis at baseline imaging
* Pancreatic surgery at baseline imaging in our department
* Splenectomy
* Patients with significant alcohol consumption, defined as alcohol intake of over 20 g daily (140 g weekly) for men and 10 g daily (70 g weekly) for women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 - pancreatic cystic neoplastic lesion Group 2 - pancreatic ductal adenocarcinoma Group 3 - control
Sampling Method: Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
increased prevalence of pancreatic steatosis in neoplastic cystic lesions | From enrollment up to 5 years
  Increased prevalence of pancreatic steatosis in neoplastic cystic lesions (mostly premalignant lesions)

SECONDARY OUTCOMES:
Increased prevalence of pancreatic steatosis in PDAC | From enrollment up to 5 years
  The investigators are looking for increased prevalence of pancreatic steatosis in patients with PDAC and its association with stage of PDAC and PDAC-related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Ciocirlan, MD PhD, Study Chair — Romanian Society of Digestive Endoscopy
Locations (1):
- Prof Dr Agrippa Ionescu; Clinical Emergency Hospital, Bucharest, Sector 1, Romania

IPD SHARING:
Plan to Share IPD: No
The study is single center therefore no IPD will be needed

REFERENCES:
- [Background] Rebours V, Gaujoux S, d'Assignies G, Sauvanet A, Ruszniewski P, Levy P, Paradis V, Bedossa P, Couvelard A. Obesity and Fatty Pancreatic Infiltration Are Risk Factors for Pancreatic Precancerous Lesions (PanIN). Clin Cancer Res. 2015 Aug 1;21(15):3522-8. doi: 10.1158/1078-0432.CCR-14-2385. Epub 2015 Feb 19. PMID 25700304
- [Background] Kashiwagi K, Seino T, Fukuhara S, Minami K, Horibe M, Iwasaki E, Takaishi H, Itoh K, Sugino Y, Inoue N, Iwao Y, Kanai T. Pancreatic Fat Content Detected by Computed Tomography and Its Significant Relationship With Intraductal Papillary Mucinous Neoplasm. Pancreas. 2018 Oct;47(9):1087-1092. doi: 10.1097/MPA.0000000000001103. PMID 30028443

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT06867172/Prot_SAP_ICF_000.pdf